CLINICAL TRIAL: NCT00004900
Title: A Phase II Pilot Study of Sequential High Dose Chemotherapy and CD 34+ Selected Stem Cell Support Without Conventional-Dose Induction Chemotherapy for Women With Metastatic Breast Cancer
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU-HAC98B2; CDR0000067579 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1689
Record Dates: First submitted 2000-03-07; First posted 2004-08-20 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Anastrozole; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: anastrozole
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus peripheral stem cell transplantation in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity and response rates to sequential high dose chemotherapy without induction chemotherapy in women with metastatic breast cancer. II. Determine the hematopoietic recovery rate in these patients after infusion of blood derived CD34+ progenitors isolated using a CD34+ affinity device for positive purification of the autograft. III. Compare response rates and duration of responses between these patients treated in this trial to patients treated in a previous trial using the same sequential high dose chemotherapy with induction conventional dose chemotherapy.

OUTLINE: Patients receive cyclophosphamide IV daily for 2 days, and etoposide IV and cisplatin IV daily for 3 days. Filgrastim (G-CSF) is administered subcutaneously twice daily beginning 24 hours after completion of chemotherapy until the last day of apheresis. Upon hematopoietic recovery, peripheral blood stem cells (PBSC) are collected over several days. Within 35 days of mobilization chemotherapy, patients receive cyclophosphamide IV, thiotepa IV, and carboplatin IV continuously on days -7 to -4, followed by a 2 day rest period. CD34+ selected PBSC are reinfused. Beginning 4 hours after reinfusion, patients receive G-CSF subcutaneously daily until hematopoietic recovery. Patients may then receive radiation therapy to sites of prior bulk disease at the discretion of the investigator. Within 30 days of hematopoietic recovery or immediately following post transplant radiation therapy, patients receive oral anastrazole daily until disease progression. Patients are followed monthly for 6 months, every 3 months for 1 year, every 4-6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed epithelial carcinoma of the breast metastatic to any organ except brain, including ipsilateral supraclavicular (not axillary) lymph nodes and chest wall No apocrine, adenocystic, squamous cell carcinoma, sarcoma, or lymphoma Measurable or evaluable disease No stage IV disease rendered nonassessable by surgery No symptomatic CNS disease Hormone receptor status: Must have biological and/or immunocytochemical receptor assays for estrogen and progesterone reported

PATIENT CHARACTERISTICS: Age: 18 to 65 Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 3.0 mg/dL SGOT no greater than 6 times upper limit of normal Renal: Not specified Cardiovascular: Ejection fraction at least 40% by MUGA No angina pectoris requiring active nitrate therapy No myocardial infarction within the past 6 months No uncontrolled congestive heart failure, uncontrolled hypertension, or major ventricular arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection or medical condition that would preclude administration of high dose therapy No other prior malignancy within the past 5 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix No uncompensated endocrine dysfunction HIV negative Hepatitis B negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior course of adjuvant therapy No other prior chemotherapy for metastatic breast cancer At least 6 months since prior adjuvant therapy No cumulative doxorubicin equivalent dose or greater than 360 mg/m2 in the adjuvant setting Endocrine therapy: Prior hormonal therapy for metastatic disease allowed Radiotherapy: Not specified Surgery: See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L. Pecora, MD, FACP, Study Chair — Hackensack University Medical Center Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Pecora AL, Lazarus HM, Stadtmauer EA, Winter J, Van Vliet A, Berry D, Gray R, Jennis A, Goldberg S, Cooper BW, Preti R. Effect of induction chemotherapy and tandem cycles of high-dose chemotherapy on outcomes in autologous stem cell transplant for metastatic breast cancer. Bone Marrow Transplant. 2001 Jun;27(12):1245-53. doi: 10.1038/sj.bmt.1703066. PMID 11548842
- [Background] Pecora A, Lazarus H, Stadtmauer E, et al.: Induction chemotherapy prior to sequential high dose chemotherapy compared to no induction increases the rate of complete response and duration of progression free survival in women with metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A-467, 1999.
- [Background] Pecora AL, Lazarus L, Kramer L, et al.: Phase II multi-institution trial of induction docetaxel and doxorubicin followed by sequential high dose chemotherapy for women with metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A-634, 1998.